CLINICAL TRIAL: NCT04574414
Title: NeuroSmog: Determining the Impact of Air Pollution on the Developing Brain
Brief Title: Determining the Impact of Air Pollution on the Developing Brain
Acronym: NeuroSmog
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jagiellonian University (Other)
Collaborators: Institute of Environmental Protection - National Research Institute (IOS-PIB) (Unknown); Foundation for Polish Science (Unknown)
Responsible Party: Principal Investigator, Marcin Szwed, Leader of the NeuroSmog consortium, Jagiellonian University
Other Study IDs: KE_24042019A
Record Dates: First submitted 2020-09-22; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Attention Deficit Hyperactivity Disorder; Attention; Executive Functioning; Social Functioning
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Social Adjustment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Attention Deficit Hyperactivity Disorder: Cases
  Interventions: Diagnostic Test: Psychological testing and MRI imaging
- Children without Attention Deficit Hyperactivity Disorder: Population controls
  Interventions: Diagnostic Test: Psychological testing and MRI imaging

INTERVENTIONS:
Diagnostic Test: Psychological testing and MRI imaging — Every child will have three sessions with psychologists and be diagnosed as having or not having ADHD.
  Every child will be invited to Krakow to undergo MRI measurements, including resting-state and event-related functional MRI, Diffusion Tensor Imaging (DTI), and T1/T2 structural MRI.

SUMMARY:
* Background: Recent studies have linked exposure to airborne particulate matter (PM) to neurodevelopmental outcomes but the findings are mixed and mechanisms are unclear. We aim to determine the impact of PM on the developing brain of schoolchildren in Poland, a European country characterized by very high levels of air pollution. The investigators aim to determine the impact of PM on the developing brain of schoolchildren in Poland, a European country characterized by very high levels of air pollution.
* Study area: 19 towns in three voivodeships (Lesser Poland, Silesian, Opole) in the southern Poland. To reduce confounding by urbanicity and at the same time, to achieve sufficient contrasts in PM levels without too high logistic costs, towns were selected by size (big and small) and by PM levels (high, medium and low).
* Design: Case-control study with 800 children recruited over two school years, with two population controls per one ADHD case. Suspected cases will be recruited in specialized facilities and presumably ADHD-free children will be recruited in primary schools.
* Exposure assessment: Poland-wide PM and other air pollutants' grids will be created for the years 2006 to 2021 using statistical models to incorporate land use data, estimates from transport models, satellite observations and air pollution measurements from Polish monitoring network. Prenatal, early-life, lifelong and concurrent exposures will be calculated.
* Psychological testing: Every child and their parents will complete a series of psychological tests and interviews that will be conducted during their three visits to the recruitment facility.
* Neuroimaging: Each participant will undergo a Magnetic Resonance Imaging (MRI) scanning session that will be performed accordingly to the Human Connectome Adolescent Brain Cognitive Development project recommendations. Scanning will be performed on a single scanner in Krakow.

ELIGIBILITY:
Inclusion Criteria:

* Attending school in one of the specified towns
* Age 10-13 years (4th-6th grade)
* Native Polish speaker
* Normal or above intelligence
* Standard educational opportunities
* Normal or corrected to normal visual and auditory acuity
* No gross sensory deficit, no gross behavioural problems
* No history of neurological disease

Exclusion Criteria:

* Autism spectrum disorder (ASD)
* FAS
* FAE
* Intellectual disability
* Metabolic disorders
* Genetic disorders
* Epilepsy
* Cerebral palsy
* Mood disorders
* Tourette Syndrome
* Other illnesses including pharmacotherapy
* Apgar score < 8
* Low birth weight (below 2500 g)
* Preterm birth (below 35th weeks of gestation)

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 800 children aged 10-13 will be sampled to the NeuroSmog study. Both ADHD cases and population controls will be enrolled, two control per case. Cases will be recruited in specialized facilities and controls will be randomly sampled in randomly selected 30 primary schools across 19 big and small towns in Lesser Poland, Silesian and Opole voivodeships in the southern Poland.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Attention Deficit Hyperactivity Disorder (ADHD) | October 1, 2020 until December 31, 2022
  ADHD and comorbidities will be assessed by Conners 3 questionnaire
Cognitive functioning | October 1, 2020 until December 31, 2022
  Memory, attention, and executive functions measurement will be assessed by Diagnostic battery for cognitive functions evaluation (PU1)
Attention control | October 1, 2020 until December 31, 2022
  Attention Network Test (ANT) will be used.
Sustained and selective attention | October 1, 2020 until December 31, 2022
  Computer Conners Continuous Performance Task (CPT) will be used.
Inhibition control | October 1, 2020 until December 31, 2022
  Conditioned Approach Response Inhibition Task (CARIT) will be used as part of MRI measurements.
Inhibition control | October 1, 2020 until December 31, 2022
  Go/No Go task will be used as part of MRI measurements.

SECONDARY OUTCOMES:
Full-Scale Intelligence Quotient (IQ) | October 1, 2020 until December 31, 2022
  IQ will be measured by Stanford-Binet Intelligence Scales, 5th Edition (SB5).
Family functioning | October 1, 2020 until December 31, 2022
  Polish adaptation of the FACES-IV (Flexibility and Cohesion Evaluation Scales; SOR) will be used to estimate social functioning of the children (family functioning).
Relationships with siblings | October 1, 2020 until December 31, 2022
  Siblings Relationship Questionnaire (KRR), which is a supplement for the SOR Scale will be used to assess social functioning of the children (relationships with siblings).
Behavioural, emotional, and social problems | October 1, 2020 until December 31, 2022
  Youth Self-Report Scale (YSR) will be used for this assessment.
Behavioural problems | October 1, 2020 until December 31, 2022
  Child Behaviour Checklist (CBCL) questionnaire will collect information on the eight syndrome domains: anxious/depressed, depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behaviour, aggressive behaviour

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychology, Krakow, Poland

REFERENCES:
- [Derived] Sitnik-Warchulska K, Izydorczyk B, Sawicki A, Markevych I, Szwed M, Lipowska M. A Dyadic Perspective on ADHD: Adolescent-Parent Reports of Behavioural Problems and Family Functioning. Clin Psychol Psychother. 2026 Jan-Feb;33(1):e70230. doi: 10.1002/cpp.70230. PMID 41603676
- [Derived] Compa M, Walczak B, Baumbach C, Kolodziejczyk J, Mysak Y, Lipowska M, Izydorczyk B, Sitnik-Warchulska K, Markevych I, Szwed M. Association of Socioeconomic Status With IQ and Attention in School Children in Poland, a Country With Relatively Low Socioeconomic Differences. Dev Psychobiol. 2025 Jul;67(4):e70058. doi: 10.1002/dev.70058. PMID 40534211